CLINICAL TRIAL: NCT06751108
Title: Impact of Concomitant Use of Steroids and Immune-Checkpoint Inhibitors on Survival Outcomes in NSCLC Patients: a Multicenter Target Trial Emulation Study Utilizing EHR-based Common Data Models
Brief Title: Impact of Concomitant Use of Steroids and Immune-Checkpoint Inhibitors on Survival Outcomes in NSCLC Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University (Other)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Pusan National University Hospital (Other); Catholic Medical Center of Korea (Unknown)
Responsible Party: Principal Investigator, Jung Mi Oh, Professor, Seoul National University
Other Study IDs: E-2024-4237
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: NSCLC, Non Small Cell Lung Cancer
Keywords: NSCLC; Non small cell lung cancer; ICI; Immune check point inhibitor; corticosteroid
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Adrenal Cortex Hormones; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Steroid Concomitant Group: Patients who received systemic corticosteroids concomitantly during the initial continuous administration period of immune checkpoint inhibitors.
  Interventions: Drug: Corticosteroids (CS); Drug: Immune Checkpoint Inhibitors
- Steroid Non-Concomitant Group: Patients who did not receive systemic corticosteroids concomitantly during the initial continuous administration period of immune checkpoint inhibitors.
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Corticosteroids (CS) — Concomitant use of immune checkpoint inhibitors and corticosteroids
  Groups: Steroid Concomitant Group
Drug: Immune Checkpoint Inhibitors — Non-concomitant use of corticosteroids

SUMMARY:
The goal of this observational study is to assess the effects of systemic corticosteroid use during immune checkpoint inhibitor (ICI) therapy in patients with non-small cell lung cancer (NSCLC). The main question it aims to answer is:

Does the use of systemic corticosteroids during the initial continuous administration of ICI therapy affect overall survival (OS) and treatment outcomes in NSCLC patients?

Participants who received ICI therapy (nivolumab, pembrolizumab, atezolizumab, or durvalumab) between December 31, 2014, and December 31, 2021, as part of their routine medical care, will be included. Patient data will be analyzed retrospectively using clinical data from five institutions, and a 1:1 propensity score matching method will be employed to balance the baseline characteristics between groups. Statistical analyses will focus on overall survival, time-to-next-treatment (TNT), and metastasis-free survival (MFS).

DETAILED DESCRIPTION:
Purposive sampling was employed to select participants who met the specific inclusion criteria, focusing on patients diagnosed with non-small cell lung cancer (NSCLC) and treated with immune checkpoint inhibitors (ICI) (nivolumab, pembrolizumab, atezolizumab, or durvalumab) during routine clinical practice. The study specifically targets patients who received their first ICI therapy between December 31, 2014, and December 31, 2021. Participants are restricted to those diagnosed with NSCLC within 2 years prior to the date of first ICI administration. Patients with documented pregnancy within 180 days prior to the enrollment date were excluded, as were those under 18 years of age or over 100 years of age at the time of enrollment. Individuals with a history of any primary malignancy other than lung cancer within 2 years prior to the enrollment date and those who received concomitant anticancer therapies such as taxane, platinum, pemetrexed, etoposide, doxorubicin, gemcitabine, irinotecan, vinorelbine, vinblastine, or bevacizumab at the index date were also excluded. All participants were identified retrospectively from clinical data models (CDM) or electronic medical records (EMRs) across five institutions: Seoul National University Hospital, Bundang Seoul National University Hospital, Pusan National University Hospital, and the Catholic Medical Center of Korea. To minimize selection bias inherent to observational studies, time-dependent propensity score matching was performed, simulating pseudo-randomization to balance baseline characteristics between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received immune checkpoint inhibitor (ICI) therapy (nivolumab, pembrolizumab, atezolizumab, or durvalumab) for the first time between December 31, 2014 and December 31, 2021.
* Patients diagnosed with non-small cell lung cancer (NSCLC) within 2 years prior to the date of first ICI administration.

Exclusion Criteria:

* Patients with documented pregnancy within 180 days prior to the enrollment date.
* Patients who were under 18 years of age or over 100 years of age at the time of enrollment.
* Patients with a history of any primary malignancy other than lung cancer within 2 years prior to the enrollment date.
* Patients who received concomitant anticancer therapies (taxane, platinum, pemetrexed, etoposide, doxorubicin, gemcitabine, irinotecan, vinorelbine, vinblastine, or bevacizumab) at the index date.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be established by constructing cohorts from patients treated at the following four hospitals: Seoul National University Hospital, Bundang Seoul National University Hospital, Pusan National University Hospital, and the Seoul Catholic Medical Center of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From index date to the end of 2 years follow-up

SECONDARY OUTCOMES:
Metastasis-free survival | From index date to the end of 2 years follow-up
  Duration of survival without distant metastasis
Time-to-next-treatment | From index date to the end of 2 years follow-up
  Time to treatment switch
Hospitalization | From index date to the end of 2 years follow-up
  Emergency room visit or hospitalization lasting more than 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This is an observational study using a common data model as the data source, where raw data at the individual patient level cannot be exported or managed externally.